CLINICAL TRIAL: NCT02681484
Title: Speech Guided Breathing: a Modality to Influence Cardiovascular Regulation and Health Perception in Hypertensive Patients?
Brief Title: Effects of Speech-therapy in Hypertensive Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Klinik Arlesheim (Other)
Collaborators: Paracelsus-Spital Richterswil (Unknown); University of Bern (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Factorial | Masking: None | Purpose: Treatment
Other Study IDs: ATS1
Record Dates: First submitted 2015-10-30; First posted 2016-02-12 (Estimated); Last update posted 2016-02-12 (Estimated); Status verified 2016-02

CONDITIONS: Hypertension
MeSH Terms: conditions — Hypertension

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Hypertensive (Experimental): Patients diagnosed with hypertension (I10, either on drug therapy or verified by 24h blood pressure measurements) administered to anthroposophic speech therapy (intervention).
  Interventions: Behavioral: Anthroposophic speech therapy
- Normotensive (Active Comparator): Patients diagnosed with tension headache (G 44.2) or anxiety disorders (F41) administered to anthroposophic speech therapy (intervention).
  Interventions: Behavioral: Anthroposophic speech therapy

INTERVENTIONS:
Behavioral: Anthroposophic speech therapy — Anthroposophic speech therapy uses sound-combinations like "KLSFM" or "OM" and hexameter verse in German, spoken by the therapist and imitated by the patients, to expand and decelerate respiration. The intervention is conducted by the same qualified therapist for one patient in different days but during the same daytime for 30 minutes in upright position and walking.
  Other Names: Speech guided breathing therapy

SUMMARY:
Anthroposophic speech therapy (ATS) has been shown to positively influence heart rate variability (HRV) and heart rate - respiration coordination in healthy volunteers. This study was performed to learn more about such improvements and possible alteration in baroreflex sensitivity (BRS) in hypertensive patients, which characteristically differ in those regulatory parameters from normotensive patients

DETAILED DESCRIPTION:
In this prospective, primarily pre-post study, patients received three ATS treatments in alternation with three control sessions (casual talking with the therapist). In order to perform HRV-analysis and BRS determination blood pressure and ECG were continuously recorded during the sessions. Changes in subjective well-being and perceived health were assessed by questionnaire before and after the various sessions (mood questionaire).

Thirty-one patients participated in this study, the majority diagnosed with arterial hypertension (22 out of 31).

ELIGIBILITY:
Inclusion Criteria:

* Indication for speech therapy
* Willing and able to perform speech therapy
* Out-patient treatment or planned hospitalisation for at least 14 days.
* Diagnosed with hypertension (I 10, either on drug therapy or verified by 24h blood pressure measurements), with tension headache (G 44.2) or with anxiety (F 41) confirmed by the recruiting physician
* No alteration in medication affecting HRV for the last 2 months before and during the study

Exclusion Criteria:

* Comorbidity strongly influencing HRV
* Too weak to participate in an active therapy
* Pacemaker
* Skin disease or allergies preventing the use of ECG electrodes

Ages: 20 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 31 (Actual)
Dates: Start 2002-09; Primary Completion 2008-04 (Actual); Study Completion 2008-04 (Actual)

PRIMARY OUTCOMES:
Change from pre-rest baroreflex sensitivity after intervention and resting. | 30min in total per session. Six sessions per patient in total.
  Baro reflex sensitivity via continuous blood pressure measurement by volume clamp method (non invasive)

SECONDARY OUTCOMES:
Change from pre-rest heart rate variability after intervention and resting | Measurement over whole session (60min in total). Six sessions per patient in total.
  Heart rate variability measurements via portable ECG-recorder

CONTACTS AND LOCATIONS:
Overall Officials: Christoph Kaufmann, PhD, Study Director — Chief Physician

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Simoes-Wust AP, Rist L, Dettling M. Self-reported health characteristics and medication consumption by CAM users and nonusers: a Swiss cross-sectional survey. J Altern Complement Med. 2014 Jan;20(1):40-7. doi: 10.1089/acm.2012.0762. Epub 2013 Jul 17. PMID 23863087
- [Background] Brook RD, Appel LJ, Rubenfire M, Ogedegbe G, Bisognano JD, Elliott WJ, Fuchs FD, Hughes JW, Lackland DT, Staffileno BA, Townsend RR, Rajagopalan S; American Heart Association Professional Education Committee of the Council for High Blood Pressure Research, Council on Cardiovascular and Stroke Nursing, Council on Epidemiology and Prevention, and Council on Nutrition, Physical Activity. Beyond medications and diet: alternative approaches to lowering blood pressure: a scientific statement from the american heart association. Hypertension. 2013 Jun;61(6):1360-83. doi: 10.1161/HYP.0b013e318293645f. Epub 2013 Apr 22. PMID 23608661
- [Background] Mancia G, Grassi G, Giannattasio C, Seravalle G. Sympathetic activation in the pathogenesis of hypertension and progression of organ damage. Hypertension. 1999 Oct;34(4 Pt 2):724-8. doi: 10.1161/01.hyp.34.4.724. PMID 10523349
- [Background] Mancia G, Grassi G. Mechanisms and clinical implications of blood pressure variability. J Cardiovasc Pharmacol. 2000;35(7 Suppl 4):S15-9. doi: 10.1097/00005344-200000004-00003. PMID 11346215
- [Background] Jonas WB. Reframing placebo in research and practice. Philos Trans R Soc Lond B Biol Sci. 2011 Jun 27;366(1572):1896-904. doi: 10.1098/rstb.2010.0405. PMID 21576147
- [Background] Bernardi L, Sleight P, Bandinelli G, Cencetti S, Fattorini L, Wdowczyc-Szulc J, Lagi A. Effect of rosary prayer and yoga mantras on autonomic cardiovascular rhythms: comparative study. BMJ. 2001 Dec 22-29;323(7327):1446-9. doi: 10.1136/bmj.323.7327.1446. PMID 11751348
- [Background] Cysarz D, von Bonin D, Brachmann P, Buetler S, Edelhauser F, Laederach-Hofmann K, Heusser P. Day-to-night time differences in the relationship between cardiorespiratory coordination and heart rate variability. Physiol Meas. 2008 Nov;29(11):1281-91. doi: 10.1088/0967-3334/29/11/004. Epub 2008 Oct 9. PMID 18843164
- [Background] von Bonin D, Grote V, Buri C, Cysarz D, Heusser P, Moser M, Wolf U, Laederach K. Adaption of cardio-respiratory balance during day-rest compared to deep sleep--an indicator for quality of life? Psychiatry Res. 2014 Nov 30;219(3):638-44. doi: 10.1016/j.psychres.2014.06.004. Epub 2014 Jun 9. PMID 25011731
- [Background] Villa MP, Calcagnini G, Pagani J, Paggi B, Massa F, Ronchetti R. Effects of sleep stage and age on short-term heart rate variability during sleep in healthy infants and children. Chest. 2000 Feb;117(2):460-6. doi: 10.1378/chest.117.2.460. PMID 10669691
- [Background] Sztajzel J. Heart rate variability: a noninvasive electrocardiographic method to measure the autonomic nervous system. Swiss Med Wkly. 2004 Sep 4;134(35-36):514-22. doi: 10.4414/smw.2004.10321. PMID 15517504
- [Background] Berntson GG, Bigger JT Jr, Eckberg DL, Grossman P, Kaufmann PG, Malik M, Nagaraja HN, Porges SW, Saul JP, Stone PH, van der Molen MW. Heart rate variability: origins, methods, and interpretive caveats. Psychophysiology. 1997 Nov;34(6):623-48. doi: 10.1111/j.1469-8986.1997.tb02140.x. PMID 9401419
- [Background] Heart rate variability. Standards of measurement, physiological interpretation, and clinical use. Task Force of the European Society of Cardiology and the North American Society of Pacing and Electrophysiology. Eur Heart J. 1996 Mar;17(3):354-81. No abstract available. PMID 8737210
- [Background] Oka H, Mochio S, Yoshioka M, Morita M, Inoue K. Evaluation of baroreflex sensitivity by the sequence method using blood pressure oscillations and R-R interval changes during deep respiration. Eur Neurol. 2003;50(4):230-43. doi: 10.1159/000073865. PMID 14634268
- [Background] Walchli C, Saltzwedel G, Kruerke D, Kaufmann C, Schnorr B, Rist L, Eberhard J, Decker M, Simoes-Wust AP. Physiologic effects of rhythmical massage: a prospective exploratory cohort study. J Altern Complement Med. 2014 Jun;20(6):507-15. doi: 10.1089/acm.2012.0833. Epub 2013 May 23. PMID 23700977
- [Background] Seifert G, Driever PH, Pretzer K, Edelhauser F, Bach S, Laue HB, Langler A, Musial-Bright L, Henze G, Cysarz D. Effects of complementary eurythmy therapy on heart rate variability. Complement Ther Med. 2009 Jun;17(3):161-7. doi: 10.1016/j.ctim.2008.09.005. Epub 2008 Nov 20. PMID 19398070
- [Background] Cysarz D, von Bonin D, Lackner H, Heusser P, Moser M, Bettermann H. Oscillations of heart rate and respiration synchronize during poetry recitation. Am J Physiol Heart Circ Physiol. 2004 Aug;287(2):H579-87. doi: 10.1152/ajpheart.01131.2003. Epub 2004 Apr 8. PMID 15072959
- [Background] Bettermann H, von Bonin D, Fruhwirth M, Cysarz D, Moser M. Effects of speech therapy with poetry on heart rate rhythmicity and cardiorespiratory coordination. Int J Cardiol. 2002 Jul;84(1):77-88. doi: 10.1016/s0167-5273(02)00137-7. PMID 12104068
- [Background] von Bonin D, Fruhwirth M, Heuser P, Moser M. [Effects of speech therapy with poetry on heart rate variability and well-being]. Forsch Komplementarmed Klass Naturheilkd. 2001 Jun;8(3):144-60. doi: 10.1159/000057212. German. PMID 11509858
- [Background] Grossman E, Grossman A, Schein MH, Zimlichman R, Gavish B. Breathing-control lowers blood pressure. J Hum Hypertens. 2001 Apr;15(4):263-9. doi: 10.1038/sj.jhh.1001147. PMID 11319675
- [Background] Moser M, Fruhwirth M, Penter R, Winker R. Why life oscillates--from a topographical towards a functional chronobiology. Cancer Causes Control. 2006 May;17(4):591-9. doi: 10.1007/s10552-006-0015-9. PMID 16596315
- [Background] Parati G, Ochoa JE, Bilo G. Blood pressure variability, cardiovascular risk, and risk for renal disease progression. Curr Hypertens Rep. 2012 Oct;14(5):421-31. doi: 10.1007/s11906-012-0290-7. PMID 22903810
- [Background] Gillette MU, Sejnowski TJ. Physiology. Biological clocks coordinately keep life on time. Science. 2005 Aug 19;309(5738):1196-8. doi: 10.1126/science.1111420. No abstract available. PMID 16109872
- [Background] Kienle GS, Albonico HU, Baars E, Hamre HJ, Zimmermann P, Kiene H. Anthroposophic medicine: an integrative medical system originating in europe. Glob Adv Health Med. 2013 Nov;2(6):20-31. doi: 10.7453/gahmj.2012.087. PMID 24416705